CLINICAL TRIAL: NCT01628510
Title: Randomized Clinical Trial Investigating the Developmental Effects of Two Different Methods of Neonatal Positioning in the NICU
Brief Title: The Developmental Effects of NICU Positioning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Roberta Pineda, Research Assistant Professor, Washington University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201111170
Record Dates: First submitted 2012-06-19; First posted 2012-06-26 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-01

CONDITIONS: Premature Birth of Newborn
Keywords: preterm
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Traditional NICU Positioning (Active Comparator): Methods of positioning in the NICU have been used for several decades. These methods aim at providing containment and flexion and may consist of interventions such as swaddling, use of boundaries around the infant, rolled blankets, Snuggly®, or Bendy Bumper® The continued use of these methods of positioning is the control group in the current study.
  Interventions: Other: Traditional NICU Positioning
- Dandle Roo/Dandle Wrap (Experimental): The new Dandle Roo and Dandle Wrap were developed by NICU professionals to support the neurodevelopment of the preterm infant, and this device is produced by Dandle Lion Medical. The Dandle Roo/Wrap provides all around contact, containment, and proprioceptive input, (which more closely mimics the uterine environment) and can decrease excitability and promote self-regulation, while also allowing for movement with recoil back to flexion.
  Interventions: Device: Dandle Roo/Dandle Wrap

INTERVENTIONS:
Device: Dandle Roo/Dandle Wrap — Infant remains in the Dandle Roo/Dandle Wrap throughout the NICU stay when the infant is lying in the isolette or crib, but is taken out for hands on care times or when held.
  Other Names: Dandle Roo; Dandle Wrap
  Arms: Dandle Roo/Dandle Wrap
Other: Traditional NICU Positioning — These methods aim at providing containment and flexion and may consist of interventions such as swaddling, use of boundaries around the infant, rolled blankets, Snuggly®, or Bendy Bumper®
  Other Names: Snuggly®; Bendy Bumper®
  Arms: Traditional NICU Positioning

SUMMARY:
The purpose of this study is to investigate the developmental effects of two different types of positioning used with premature infants in the neonatal intensive care unit.

DETAILED DESCRIPTION:
Infants born prematurely have a high risk of developmental impairment. Subsequently, preterm infants are often seen by therapy services in the neonatal intensive care unit and are often recommended for early intervention services at discharge. One of the earliest interventions for preterm infants in the Neonatal Intensive Care Unit (NICU) is positioning, as altered positioning can have a significant impact on later function.

Preterm infants have a positioning disadvantage from early on in their development. The final trimester of pregnancy promotes the flexed position, when the infant is crowded by the uterine environment and experiences rapid brain growth, mediating flexion and midline orientation. When infants are born too soon, they miss the in utero flexion positioning. They lack the central nervous system maturity to enable flexion and do not have the tone and strength for movement against gravity. In addition, preterm infants are confronted with altered sensory experiences, resulting from static, extended positioning and environmental factors associated with life and medical interventions outside the womb. Therefore, early transition to the extrauterine environment is a challenge for premature infants, as they face overwhelming sensory stimuli that their bodies are not yet prepared to process.

It has been demonstrated that the positioning of the preterm infant differs from that of a full term infant. The tightly flexed positioning of a full term newborn is called physiological flexion. It involves symmetrical flexion of the extremities, shoulder protraction, and posterior pelvic tilt.

Physiological flexion has developmental importance. This positioning enables infants to remain motorically and physiologically organized and facilitates self-soothing and self-regulation behaviors, such as sucking and hand to mouth contact. The flexed position provides the infant with a sense of containment and security, which mimics the intrauterine environment. In addition, physiological flexion is associated with greater extremity contact with the trunk, which imitates the womb and gives infants sensory feedback.

The benefits of early physiological flexion can have long term benefits on development. Many neonatal reflexes, such as upper and lower extremity recoil, palmar and plantar grasp, and pull to sit are mediated by flexion response. These early flexion responses form the foundation for later movement acquisition. Physiological flexion also promotes later development of normal balance and posture. Ideal posture supports the development of head control, sitting, crawling, walking, transferring from one position to another, and manipulating objects. Due to missing the third trimester, preterm infants are at risk for assuming suboptimal positions, thus missing the early benefits of physiological flexion.

In utero, fetuses experience attenuated stimuli. Therefore, sensory experiences outside the womb are overwhelming for infants born prematurely (3). As a result, preterm infants are easily stressed, particularly when they are not properly positioned.

Stress can produce severe consequences in the preterm infant including respiratory problems and intraventricular hemorrhage. Infants in an unsupported position may have frantic movements and startles in response to stress, and therefore have difficulty achieving the deep sleep state necessary for growth and brain development. This can lead to extended hospital stays. Optimal positioning enables premature infants to better cope with stressors and bring their hand to face and mouth for self-soothing.

Positioning aids in the past have aimed at promoting containment and increasing flexion. However, the ability to promote flexion while enabling infant movement remained problematic. The new Dandle Roo and Dandle Wrap were developed by NICU professionals to support the neurodevelopment of the preterm infant. The Dandle Roo/Wrap provides all around contact, containment, and proprioceptive input, (which more closely mimics the uterine environment) and can decrease excitability and promote self-regulation, while also allowing for movement with recoil back to flexion.

Despite the current evidence on effective positioning interventions for preterm infants, a recent meta-analysis on developmental care cited a need for more research of specific interventions, such as positioning, on short-term and long-term clinical outcomes. No studies to date have examined the effects of the new Dandle Roo and Dandle Wrap on clinical and neurobehavioral outcomes in preterm infants. Therefore, we propose a randomized controlled trial of the new Dandle Roo/ Dandle Wrap, postulating that infants positioned in the Dandle Roo/Dandle Wrap will experience beneficial effects.

Objectives:

Hypothesis - Preterm infants positioned in the Dandle Roo and Dandle Wrap will experience better neurodevelopmental outcome, less brain injury and need for respiratory support, and shorter hospital stays than infants positioned in traditional NICU positioning aids.

Specific Aim - To conduct a randomized controlled trial on the effects of the Dandle Roo/Dandle Wrap versus traditional NICU positioning administered from birth through discharge from the NICU on neurodevelopmental outcome, brain injury, need for respiratory support, and length of stay in infants born less than 32 weeks postmenstrual age (PMA).

Subjects: A power analysis revealed that 86 infants were needed to detect a difference in neurobehavioral outcome following a positioning intervention. To account for attrition, 100 infants will be recruited.

Inclusion Criteria - This is a prospective cohort with premature infants who are born at 32 weeks or less PMA. This cohort will be hospitalized in the NICU at St. Louis Children's Hospital or the Barnes Special Care Nursery in St. Louis, Missouri and will be recruited within 72 hours of birth.

Exclusion Criteria - Infants with a known or suspected congenital anomaly at birth and infants who are moribund with severe sepsis or respiratory distress defined as physiologic instability requiring >80% FiO2 for 6 hours and/or more than 2 ionotropic drugs (excluding hydrocortisone), or in the attending or recruiting physicians' opinion the infant is likely to expire within 24 hours or would not tolerate any handling for the protocol

Randomization - As soon after birth as possible, but no later than 1 week after admission, consecutive new admissions meeting the inclusion criteria will be recruited for the study. Upon parent's signing the informed consent, an infant will be randomly assigned to either Dandle Roo/Dandle Wrap positioning or to traditional NICU positioning for the entire length of stay.

The positioning protocol assigned to each study infant would be clearly posted at each infant's bedside. Members of the research team would routinely check in to ensure that infants in the treatment arm were positioned correctly in the Dandle Roo/Dandle Wrap and to answer any questions. In addition, a log sheet would be placed at the infant's bedspace for each nursing shift. Here nurses would be instructed to identify if the infant was positioned in the assigned positioning aid and would be able to identify reasoning if the positioning was not implemented during a specific shift.

Positioning protocols would be utilized during times when the infant is resting in the crib, isolette, or open warmer. However, the infant would be taken out of the positioning aids periodically for hands on care, for bedside evaluation, or to enable closer observation during acute episodes. In addition, parents could take the infant out of the positioning for holding and interaction.

Clinical Data Collection:

For all infants enrolled, routine clinical information from the infant's medical record would be accessed.

In addition, each infant would undergo neurobehavioral testing by a member of the research team during the hospitalization. One trained and certified evaluator will conduct all neurobehavioral tests on all study infants. Testing would be conducted between 35 weeks gestation and 41 weeks gestation. Neurobehavioral assessment that will be used is the Neonatal NICU Network Scales (NNNS). Scores range from 0-13 in the following subscales: habituation, attention, handling, arousal, regulation, quality of movement, reflexes, asymmetrical responses, hypertonicity, hypotonicity, stress/abstinence signs. High scores are optimal on the following subscales: habituation, attention, regulation, and quality of movement. Low scores are optimal on the following subscales: handling, arousal, reflexes, asymmetrical responses, hypertonicity, hypotonicity and stress/abstinence signs.

Developmental testing would only be conducted on infants who were medically stable and able to tolerate the exam. Video taping of each neurobehavioral assessment will be performed and stored anonymously. Videotapes will be conducted to enable close observation of the infant during the evaluation process with later scoring of the test from the videotape. In addition, testing from the ongoing developmental follow up clinic (Washington University Neonatal Developmental Follow-Up Clinic) would be accessed for outcomes at 6 months, 1 year, 2 years, and 3 years, when available.

Dissemination of results:

The findings from this research will be:

* Published in peer review scientific medical literature
* Presented at local and international conferences
* Disseminated, at the end of the study period, to all parents whose infants were enrolled in the study who expressed interest in the study outcome.

Potential Benefits:

Ideal neonatal positioning may improve neurodevelopment and decrease brain injury and need for respiratory support, with subsequent better developmental outcome. Optimizing positioning and facilitating more optimal in utero positioning during this time period could result in shorter hospital stays, decreasing expenditure of healthcare dollars. Early neurobehavioral testing, which is part of the study protocol, can enable parents to better understand the strengths and weaknesses exhibited by their infant to enable early therapeutic interventions. Benefits to society include a better understanding of effective positioning in the NICU as well as a possible understanding about how early positioning can be critical for later function.

A member of the research team will conduct a comprehensive developmental test on the infant during the NICU stay. Parents will be informed of test results prior to or at NICU discharge.

The WUNDER research group will be continuously reviewing the data results as they return and report any adverse effects monthly to the St. Louis Children's Hospital Neonatal Intensive Care Unit Joint Practice Committee. The biostatistician will also independently review data results and report any significant adverse effects monthly to the WUNDER research group and the Joint Practice Committee. All serious adverse events will be reported to the IRB: a) death - immediately; b) life-threatening within 7 calendar days; c) all other significant adverse events (SAEs) within 15 calendar days using the Electronic SAE System.

Data Analysis:

Data will be analyzed using linear and logistic regression models by a biostatistician. Data will be reviewed throughout the duration of the study. All data will be maintained in the strictest confidence and will only be available to members of the research team. It will be held in secure format in password-protected computer records. Hard copy and the records will be identified only by study number and stored in a locked file cabinet. A log of study number and identifying data will be kept by the site PI in a separate locked file cabinet. All file cabinets containing data are inside a locked office in a corridor accessible only with badge access.

ELIGIBILITY:
Inclusion Criteria:Inclusion:

* Premature infants born at or before 32 weeks gestation

Exclusion Criteria:

* Congenital Anomaly

Ages: 1 Hour to 7 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2011-01; Primary Completion 2011-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roberta G Pineda, PhD OTR/L, Principal Investigator — Washington University School of Medicine
Locations (2):
- United States (2):
  - Barnes Special Care Nursery, St Louis, Missouri
  - St Louis Children's Hospital, St Louis, Missouri

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One hundred infants were enrolled from January 2011 through November 2011. Four infants withdrew, and four infants died. Ninety two participants were discharged from the NICU.
Pre-assignment Details: All eligible infants were recruited. Those whose parents signed informed consent were randomized to either traditional positioning or Dandle Roo positioning.
Groups:
- Traditional NICU Positioning: Methods of positioning in the NICU have been used for several decades. These methods aim at providing containment and flexion and may consist of swaddling, use of boundaries around the infant, rolled blankets, Snuggly®, or Bendy Bumper® The continued use of these methods of positioning is the control group in the current study.
Period: Overall Study
Arm/Group | Dandle Roo/Dandle Wrap | Traditional NICU Positioning
Started | 51 | 49
Completed | 48 | 44
Not Completed | 3 | 5
Not completed — Withdrawal by Subject | 0 | 4
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Traditional NICU Positioning: Methods of positioning in the NICU have been used for several decades. These methods aim at providing containment and flexion and may consist of swaddling, use of boundaries around the infant, rolled blankets, Snuggly®, or Bendy Bumper® The continued use of these methods of positioning is the control group in the current study.
  Traditional Positioning: Traditional positioning methods are used with the infant throughout the NICU hospitalization.
- Dandle Roo/Dandle Wrap: The new Dandle Roo and Dandle Wrap were developed by NICU professionals to support the neurodevelopment of the preterm infant, and this device is produced by Dandle Lion Medical. The Dandle Roo/Wrap provides all around contact, containment, and proprioceptive input, (which more closely mimics the uterine environment) and can decrease excitability and promote self-regulation, while also allowing for movement with recoil back to flexion.
  Dandle Roo/Dandle Wrap: Infant remains in the Dandle Roo/Dandle Wrap throughout the NICU stay when teh infant is lying in the isolette or crib, but is taken out for hands on care times or when held.
- Total: Total of all reporting groups
Arm/Group | Traditional NICU Positioning | Dandle Roo/Dandle Wrap | Total
Number analyzed (Participants) | 44 | 48 | 92
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 29.4 (2.8) | 28 (2.5) | 28.7 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 26 | 53
  Male | 17 | 22 | 39

OUTCOME MEASURES:

1. Primary Outcome: NICU Network Neurobehavioral Scale (NNNS)
Description: The NNNS wasl used to assess neurobehavioral outcome near term equivalent (between 35 weeks and 41 weeks postmenstrual age). This tool consists of eliciting neonatal reflexes and observing behavior. From the assessment, 13 summary scores were determined for each of the following constructs: habituation (1-9), orientation (1-9), self regulation (1-9), tolerance of handling (0-1), hypertonia (0-10), hypotonia (0-10), asymmetry (0-16), lethargy (0-15), excitability (0-15), sub-optimal reflexes (0-15), arousal (1-9), quality of movement (1-9) and stress (0-1). Each summary score is analyzed for associations with subsequent developmental outcome. A higher score in each category indicates more of that construct. Specifically, for the summary score of asymmetry (the significant finding in this study), higher scores equal more asymmetry.
Time Frame: 35 to 41 weeks (term equivalent); prior to NICU discharge
Measure: Mean (Standard Deviation); unit: Asymmetry Score (units on a scale)
Arm/Group | Traditional NICU Positioning | Dandle Roo/Dandle Wrap
Number analyzed (Participants) | 44 | 48
Asymmetry Score (units on a scale) | 3.1 (2.1) | 2.56 (1.9)

2. Secondary Outcome: The Bayley Scales of Infant Development-3rd Edition (BSID-III)
Description: The BSID-III is the gold standard for assessing developmental outcome in childhood. Subscale composite scores for language, motor and cognition will be determined.
  * Language
    --Scale Range (higher values represent a better outcome)
    * Minimum Score: 40
    * Maximum Score: 160
  * Motor
    --Scale Range (higher values represent a better outcome)
    * Minimum Score: 40
    * Maximum Score: 160
  * Cognition --Scale Range (higher values represent a better outcome)
    * Minimum Score: 40
    * Maximum Score: 160
Time Frame: 1 year, 2 years
Population: 23 total participants completed Bayley Scales follow-up testing at 1 year; 7 total participants completed Bayley Scales follow-up testing at 2 years.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Traditional NICU Positioning | Dandle Roo/Dandle Wrap
Number analyzed (Participants) | 8 | 15
units on a scale
  Cognitive - 1 year | 90 (22.99) | 105.71 (16.97)
  Language - 1 year | 85.57 (18.93) | 94.73 (19.18)
  Motor - 1 year | 82.88 (25.27) | 96.50 (11.02)
  Cognitive - 2 year: number analyzed (Participants) | 3 | 4
  Cognitive - 2 year | 75 (8.66) | 95 (5)
  Language - 2 year: number analyzed (Participants) | 3 | 4
  Language - 2 year | 77.33 (8.5) | 91.33 (8.5)
  Motor - 2 year: number analyzed (Participants) | 3 | 4
  Motor - 2 year | 79 (13.75) | 91 (12)

ADVERSE EVENTS:
Arm/Group | Dandle Roo/Dandle Wrap | Traditional NICU Positioning
All-Cause Mortality (participants affected / at risk) | 0/48 | 0/44
Serious Adverse Events (participants affected / at risk) | 0/48 | 0/44
Other Adverse Events (participants affected / at risk) | 0/48 | 0/44

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No